CLINICAL TRIAL: NCT06425315
Title: Does Targeted Management of Undernutrition in Oncogeriatric Patients Aged 70 and Over, Undergoing Cancer Treatment and Hospitalized From January 2022 to December 2023, Improve Their Nutritional and Functional Status?
Brief Title: Management of Malnutrition in Oncogeriatrics
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_5390
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Undernutrition; Cancer
Keywords: Malnutrition; Geriartric oncology; Aged; Antineoplastic agents; Muscle strenght
MeSH Terms: conditions — Malnutrition; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncogeriatric patients with undernutrition: Our study population consists of oncogeriatric patients aged 70 and over, hospitalized in the oncogeriatric follow-up and referral unit (USSROG), with a diagnosis of moderate or severe undernutrition and undergoing cancer treatment. Patients will be recruited between January 1, 2022 and December 31, 2023.
  We anticipate a sample size of between 100 and 120 patients over this period.

SUMMARY:
In France, undernutrition affects almost three million people, a third of whom are over 70 (Diagnosing undernutrition earlier in the elderly aged 70 and over, n.d.). In fact, 30 to 70% of hospitalized elderly patients suffer from protein-energy undernutrition (denutrition_personne_agee_2007_-_recommandations.pdf, n.d.).

The Nutricancer 2 study published in 2014, demonstrated that undernutrition is common among cancer patients. Indeed, 39% of patients suffer from undernutrition and its prevalence depends on the type of cancer, with a predominance of esophagus, stomach and pancreas (60% to 66%), colon/rectum, ovary/uterus and lung (39% to 45%), hematological malignancies (34%), as well as prostate and breast (13% to 20%) (Hébuterne et al., 2014). Moreover, over the past 30 years, undernutrition has been observed in 30% to 50% of the population at the time of diagnosis and before the start of cancer treatment (Boranian et al., n. d.).

Undernutrition is often associated with several terms such as malnutrition, anorexia, sarcopenia or cachexia, which refer to geriatric or metabolic syndromes of multifactorial origin that sometimes overlap, and are often observed in cancer patients. Cancer cachexia is a metabolic syndrome associated with undernutrition of multifactorial origin (Boranian et al., n.d.). Its prevalence is around 50% to 80% in cancer patients and is an independent indicator of morbidity and mortality in this population (Nicolini et al., 2013).

Undernutrition is a major health issue in elderly cancer patients. It is therefore crucial to diagnose it early, given its high prevalence in this population and the serious complications it can lead to. In 2021, the HAS updated its recommendations on the diagnosis of undernutrition in the elderly. The diagnosis of severe undernutrition is based on several criteria, including serum albumin levels. This is a commonly used marker of nutritional status, especially in patients with involuntary weight loss. However, it is important to note that hypoalbuminemia can be observed in many pathological conditions, including inflammatory syndromes common in cancer. Therefore, interpretation of albuminemia results must take into account the patient's inflammatory status, assessed by C-reactive protein. This analysis makes it possible to distinguish undernutrition due to insufficient food intake from that associated with an inflammatory syndrome and hypercatabolism (Patry & Raynaud-Simon, 2010).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 and over with a diagnosis of moderate or severe undernutrition
* All patients with diagnosed cancer and ongoing cancer treatment.

Exclusion Criteria:

* Patients under 70 years of age
* Hospitalized patients no longer undergoing anticancer treatment
* All patients undergoing pre-habilitation for surgery

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The population of this study will be made up of oncogeriatric patients aged 70 and over, hospitalized in the USSROG unit with a diagnosis of undernutrition and undergoing anticancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-24 (Estimated)

PRIMARY OUTCOMES:
The criterion chosen to demonstrate this is: absolute albumin values in g/l in patients with moderate undernutrition and in those with severe undernutrition after the first month of hospitalization, at 2 months and then at 3 months. | It will be measured at the start of hospitalization and after the first month, at 2 months and then at 3 months.
  the variation in albumin values associated with CRP values will be collected on admission and after the first month, at 2 months and then at 3 months of hospitalization.
  These values will then be analyzed using statistical analysis software, to determine whether the results obtained are relevant and favor an improvement in albumin levels, and consequently in the patient's nutritional status.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pierre Garraud, Lyon, France

IPD SHARING:
Plan to Share IPD: No